CLINICAL TRIAL: NCT03396016
Title: Plasmatic Factor V as a Predictor of Graft Dysfunction After Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 17-6090
Record Dates: First submitted 2017-12-27; First posted 2018-01-10 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Liver Transplant Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Factor V: liver transplant patients having Factor V levels measured during their first postoperative week.

SUMMARY:
Factor V is a coagulation cofactor that is primarily produced by the liver. Previous data has suggested a correlation between factor V levels and graft dysfunction. The investigators hypothesize that Factor V may be a reliable biomarker for hepatic function after LT. Therefore, the aim of this study is to validate the use of Factor V as a predictor of graft dysfunction after LT. This is a single-center prospective validation study. Patients undergoing LT at the University Health Network will have plasmatic Factor V levels measured during postoperative week 1. Patients will be followed up to 12 months. The study outcomes will be early graft dysfunction, and graft and patient survival. Graft loss will be defined as need for retransplantation in the study period.

DETAILED DESCRIPTION:
There is no widely accepted biomarker to assess hepatic function after Liver Transplantation (LT). Factor V is a coagulation cofactor that is primarily produced by the liver. Factor V has a short half-life and its production does not depend on vitamin K, relying mainly on liver function. These singular characteristics make Factor V plasmatic levels strictly linked to liver function. Previous data has suggested a correlation between factor V levels and graft dysfunction. The investigators hypothesize that Factor V may predict graft dysfunction after LT, and become a reliable biomarker for hepatic function after LT. Therefore, the aim is to validate the use of Factor V as a predictor of graft dysfunction after LT. This is a single-center prospective validation study. Participants (patients undergoing LT at the University Health Network) will have plasmatic Factor V levels measured on postoperative days (POD) 1º, 2º, 3º, 5º and 7º. Participants will be followed up to 12 months. The study primary outcome will be early graft dysfunction as defined by Olthoff et al. Secondary outcomes will be 3-, 6- and 12-months graft and patient survival. Graft loss will be defined as need for retransplantation in the study period. Potential confounders will be assessed in a multivariate regression model. No other intervention will be done to the patients. The results of this study may validate the use of this biomarker for graft dysfunction and mortality after LT. These results will impact LT research and direct patient care.

ELIGIBILITY:
Inclusion Criteria:

* Listed for a deceased donor liver transplant at University Health Network
* Able and willing to provide informed consent

Exclusion Criteria:

* Patients unable to provide informed consent
* Recipients of live donor liver transplantation
* Re-transplants
* Recipients of multiple organs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients awaiting a liver transplantation at University Health Network
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Factor V plasma level | day 1
  Factor V plasma level
Factor V plasma level | day 3
  Factor V plasma level
Factor V plasma level | Day 5
  Factor V plasma level

SECONDARY OUTCOMES:
Graft survival | 3 months
  graft survival
Graft survival | 6 months
  graft survival
Graft survival | 12 months
  graft survival
Patient survival | 3 months
  patient survival
Patient survival | 6 months
  patient survival
Patient survival | 12 months
  patient survival

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Sapisochin, MD, Principal Investigator — Surgical staff
Locations (1):
- Toronto General Hospital (University Health Network), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No